CLINICAL TRIAL: NCT00000837
Title: Phase I/II Study of the Safety and Immunogenicity of Live-Attenuated Varicella Vaccine (Varivax) in HIV-Infected Children
Brief Title: A Study of the Safety and Effectiveness of a Chickenpox Vaccine in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: PACTG 265; 10613 (Registry Identifier: DAIDS ES Registry Number); ACTG 265
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Herpesvirus 3, Human; Viral Vaccines; AIDS-Related Complex; Vaccines, Attenuated; Chickenpox; Chickenpox Vaccine
MeSH Terms: conditions — HIV Infections; Chickenpox; AIDS-Related Complex | interventions — Herpes Zoster Vaccine

INTERVENTIONS:
Biological: Varicella Virus Vaccine (Live)

SUMMARY:
The purpose of this study is to see if it is safe to give Varivax to HIV-positive children and whether it protects children from infection. Varivax is a vaccine against varicella zoster virus (VZV), the virus that causes chickenpox (varicella) and shingles (zoster).

VZV can cause many serious complications in HIV-infected children. Varivax is a VZV vaccine that has been approved for use in healthy children. More research is needed to find out how this vaccine will affect HIV-infected children.

DETAILED DESCRIPTION:
Primary varicella infection, or chickenpox, can be devastating to HIV-infected children because complications occur at higher rates in immunocompromised hosts. Current passive prophylaxis measures with varicella-zoster immune globulin are suboptimal because administration must be repeated for each exposure during the child's lifetime and timely notification of exposure is not always possible. Since Varivax has been licensed for routine vaccination of healthy individuals, it must be determined whether this vaccine can be safely administered to HIV-infected children.

Thirty-six children who are varicella zoster virus (VZV)-naive (treatment group) receive Varivax at Weeks 0 and 12, with a possible boost at Week 52 if the patient is still seronegative for VZV and cytomegalovirus infection. Twenty children who have a history of wild-type varicella exposure within the past year (control group) receive no study treatment. All patients are either asymptomatic or mildly symptomatic for HIV infection. Patients make 12-14 visits to the clinic. [AS PER AMENDMENT 9/9/99: This study has been reorganized into two cohorts (asymptomatic and symptomatic). In the asymptomatic cohort, accrual has been completed with 40 patients in Treatment Group I and 19 in the control group. This phase of the study demonstrated that Varivax was well tolerated in 48 HIV-infected children with asymptomatic disease. The symptomatic cohort includes Treatment Groups II and III, each with 30 patients. The first 10 patients from Group II are monitored for 42 days following the first dose of vaccine before the remaining 20 are accrued. Once the first 10 patients in Group II have been evaluated with acceptable toxicity and immunologic profiles, the remaining 20 Group II and the first 10 Group III patients are enrolled. The first 10 Group III patients are also followed for acceptable toxicity and immunologic response before accrual of the remaining 20 Group III patients.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive with no symptoms or moderate symptoms.
* Are between 1 and 8 years old (consent of parent or guardian required).
* Have had a CD4 cell count greater than 200 for the past 3 months. If a child had a lower CD4 count before this time, then he/she must have been on stable anti-HIV therapy for the past 3 months.

Exclusion Criteria

Children will not be eligible for this study if they:

* Have had an infection or a fever of 101 F or higher in the past 3 days.
* Have had chickenpox or shingles. (This study has been changed. Children who had VZV infections were eligible originally.)
* Have been exposed to chickenpox or shingles in the past 4 weeks.
* Live with someone who is HIV-positive or who has a lowered immune system.
* Have certain serious diseases including tuberculosis or a disease of the immune system (other than HIV infection).
* Are allergic to any part of the chickenpox vaccine, including neomycin.
* Have recently had certain treatments or might be taking certain treatments during the study such as aspirin, VZIG, IVIG, other vaccines, steroids, anti-herpes medications, blood products, or drugs that might interfere with the immune system.

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 127
Dates: Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myron J Levin, Study Chair; Anne A Gershon, Study Chair
Locations (25):
- United States (25):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Children's Hosp. of Orange County, Orange, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - The Children's Hosp. (Univ. of Colorado, Denver) P7001 CRS, Aurora, Colorado
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - South Florida CDTC Ft Lauderdale NICHD CRS, Fort Lauderdale, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - NJ Med. School CRS, Newark, New Jersey
  - Nyu Ny Nichd Crs, New York, New York
  - Metropolitan Hosp. Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Levin MJ, Gershon AA, Weinberg A, Blanchard S, Nowak B, Palumbo P, Chan CY; AIDS Clinical Trials Group 265 Team. Immunization of HIV-infected children with varicella vaccine. J Pediatr. 2001 Aug;139(2):305-10. doi: 10.1067/mpd.2001.115972. PMID 11487761